CLINICAL TRIAL: NCT06303154
Title: Evaluation of the Performance and Safety of Mobiderm Intimate Bra in the Management of Breast Edema Related to Breast Cancer Treatment - A Prospective, Exploratory, Monocentric, Uncontrolled Clinical Study
Brief Title: Evaluation of Mobiderm Intimate Bra in the Management of Breast Edema Related to Breast Cancer Treatment
Acronym: MOBIBRA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Thuasne (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC45 MOBIBRA; ID-RCB (Other: 2023-A01937-38)
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer Surgery
Keywords: Breast cancer; Surgery; Compressive bra; Breast edema
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Prospective, exploratory, monocentric, uncontrolled clinical study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Mobiderm Intimate Bra group (Experimental): All the patients will wear MOBIDERM Intimate bra composed of a bra and a MOBIDERM pad
  Interventions: Device: Mobiderm Intimate Bra group

INTERVENTIONS:
Device: Mobiderm Intimate Bra group — At the conclusion of the surgical operation, MOBIDERM Intimate bra will be placed on the patient by the medical team. It will be recommended for the patients to wear MOBIDERM Intimate Bra during day and night for 3 weeks after the surgery, and as much time as the patients tolerate the device during the rest of the study, until 6 months after radiotherapy

SUMMARY:
The aim of this exploratory study is to assess the performance and tolerability of the MOBIDERM Intimate Bra in the management of breast edema related to breast cancer treatment.

DETAILED DESCRIPTION:
Breast cancer is the most common malignancy in women in the Western World. BCS followed by radiotherapy is a safe and effective procedure to treat patients with early-stage [Verbelen H., 2021]. But some patients are troubled by breast edema in the operated and irradiated breast. The consequences of breast edema can be : an increase in breast volume, orange peel skin, heaviness of the breast, redness of the skin, breast pain, thickening of the skin, hyperpigmented skin pores [Verbelen H., 2014]. Breast edema can also imply deterioration in patients' quality of life, physical functioning, and body image [Young-Afat D. A., 2019].

According to the literature, only a few clinical studies evaluated the value of compression medical devices in the management of breast edema.

The aim of the study is to perform a prospective, exploratory, monocentric, uncontrolled clinical study to look at the performance and safety of Mobiderm Intimate Bra in the management of breast edema related to breast cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

* Females aged 18 years and older.
* Patients who have undergone conserving surgery for breast cancer.
* Patients scheduled to undergo radiation treatment of the breast/chest wall within the next 12 weeks after surgery.
* Patients with a morphology compatible with the proposed sizes of the devices, including bust girth and cup size.
* Patients who have signed an informed consent form prior to any study intervention.
* Patients with full legal capacity and enrolled in a social security system or covered by a similar health insurance.

Exclusion Criteria:

* Patients with an A cup bra size.
* Patients with infected or acutely inflammatory skin on the chest.
* Patients who require chemotherapy during the follow-up period.
* Pregnant women or women of childbearing age without adequate contraception or in the lactation period.
* Participation in other clinical trials that impact the primary endpoint.
* Patients with a known allergy to the investigational device components.
* Patients with psychiatric, psychological, or neurological disorders that are incompatible with the conduct of a clinical trial.
* Patients unable to be followed for 12 months.
* Vulnerable patients, or those subject to a judicial protection measure or unable to provide informed consent freely.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-21 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Evolution of breast edema severity | Between 35 and 44 weeks (6 months after radiotherapy)
  The evolution of breast edema severity will be assessed all along the study follow-up using the patient-completed "Symptoms" section of the Breast Edema Questionnaire (BrEQ): 8 questions about symptoms of breast edema scored on a scale from 0 to 10 (0 = no difficulty and 10: maximal difficulty). The maximum score is 80 .

SECONDARY OUTCOMES:
Comparison of methods to follow changes in the severity of breast edema - TDC measurement | Between 35 and 44 weeks (from inclusion to 6 months after radiotherapy)
  Measurement of the Tissue Dielectric Constant (TDC) of the breast tissue will be done using the MoistureMeter D (Delfin Technologies Ltd, Finland).
Comparison of methods to follow changes in the severity of breast edema - Clinical assessment | Between 35 and 44 weeks (from inclusion to 6 months after radiotherapy)
  Clinical assessment will be done by observation and palpation of the breast by the medical team to monitor changes in the severity of breast edema.
Comparison of methods to follow changes in the severity of breast edema - Ultrasound measurement | Between 35 and 44 weeks (from inclusion to 6 months after radiotherapy)
  High-frequency cutaneous ultrasound measurements will be done by the medical team to monitor changes in the severity of breast edema (echogenicity, skin thickness).
Time to edema onset | Between 35 and 44 weeks (from inclusion to 6 months after radiotherapy)
  The time between surgery and/or radiotherapy and the diagnosis of breast edema will be assessed by analysing the responses to the "Symptoms" section of the BrEQ questionnaire completed weekly.
Time to edema disappearance | Between 35 and 44 weeks (from inclusion to 6 months after radiotherapy)
  The time to disappearance of the breast edema will be assessed by analysing the responses to the "Symptoms" section of the BrEQ questionnaire completed weekly.
Symptoms and quality of life changes associated with breast edema | Between 35 and 44 weeks (from inclusion to 6 months after radiotherapy)
  Changes in symptoms (pain, heaviness, swelling, tension, hardness and redness of the skin, etc.) and quality of life related to breast edema will be assessed by the patient by filling in the BrEQ self-questionnaire. The 8 questions related to symptoms and 16 questions related to quality of life are scored on a scale from 0 to 10 (0 = no difficulty and 10: maximal difficulty). The maximum score is 80 for the symptoms part and 160 for the Quality of life part.
Breast edema hypersensitivity | Between 35 and 44 weeks (from inclusion to 6 months after radiotherapy)
  The evolution of breast hypersensitivity will be assessed using a Visual Analogue Scale (VAS) (score from 0 to 10 with 0 = no hypersensibility and 10 = maximum hypersensibility).
Breast pain | Between 35 and 44 weeks (from inclusion to 6 months after radiotherapy)
  The presence of breast pain will be assessed using a VAS (score from 0 to 10 with 0 = no pain and 10 = Maximal pain).
Skin changes associated with breast edema | Between 35 and 44 weeks (from inclusion to 6 months after radiotherapy)
  Changes in skin fibrosis/hardness will be assessed using the SkinFibroMeter (Delfin Technologies Ltd, Finland).
Physical activity | Between 35 and 44 weeks (from inclusion to 6 months after radiotherapy)
  The time taken to resume physical activity will be measured by means of a specific question to the patient.
Healing time | Between 35 and 44 weeks (from inclusion to 6 months after radiotherapy)
  The healing time will be calculated following observation of scar oozing by the medical team.
Safety of the device | Between 35 and 44 weeks (from inclusion to 6 months after radiotherapy)
  The safety of the device will be assessed by describing the adverse events (AEs) and serious adverse events (SAEs) that occur throughout the study.
Compliance to the device | Between 35 and 44 weeks (from inclusion to 6 months after radiotherapy)
  The Investigator will report compliance with the device at each visit using the patient's diary, which the patient shall complete throughout the follow-up period
Patient's satisfaction | 3 weeks after surgery and 6 months after radiotherapy (end of study)
  Patient's satisfaction with the MOBIDERM Intimate Bra device will be evaluated with a specific self-questionnaire given to the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Séverine ALRAN, Dr, Principal Investigator — Groupe Hospitalier Paris Saint Joseph - Groupement FEHAP
Locations (1):
- Groupe Hospitalier Paris Saint Joseph - Groupement FEHAP, Paris, Paris 14, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Johansson K. et al. Two-year follow-up of temporal changes of breast edema after breast cancer treatment with surgery and radiation evaluated by tissue dielectric constant (TDC). The European Journal of Lymphology and related problem. 2015; 27:73.
- [Background] Young-Afat DA, Gregorowitsch ML, van den Bongard DH, Burgmans I, van der Pol CC, Witkamp AJ, Bijlsma RM, Koelemij R, Schoenmaeckers EJ, Jonasse Y, van Gils CH, Verkooijen HM. Breast Edema Following Breast-Conserving Surgery and Radiotherapy: Patient-Reported Prevalence, Determinants, and Effect on Health-Related Quality of Life. JNCI Cancer Spectr. 2019 Apr 16;3(2):pkz011. doi: 10.1093/jncics/pkz011. eCollection 2019 Jun. PMID 31360894
- [Background] Verbelen H, Gebruers N, Beyers T, De Monie AC, Tjalma W. Breast edema in breast cancer patients following breast-conserving surgery and radiotherapy: a systematic review. Breast Cancer Res Treat. 2014 Oct;147(3):463-71. doi: 10.1007/s10549-014-3110-8. Epub 2014 Aug 28. PMID 25164973
- [Background] Verbelen H, Tjalma W, Dombrecht D, Gebruers N. Breast edema, from diagnosis to treatment: state of the art. Arch Physiother. 2021 Mar 29;11(1):8. doi: 10.1186/s40945-021-00103-4. PMID 33775252
- [Background] Johansson K, Jonsson C, Bjork-Eriksson T. Compression Treatment of Breast Edema: A Randomized Controlled Pilot Study. Lymphat Res Biol. 2020 Apr;18(2):129-135. doi: 10.1089/lrb.2018.0064. Epub 2019 Jun 24. PMID 31233373
- [Background] Gregorowitsch ML, Van den Bongard DHJG, Batenburg MCT, Traa-van de Grootevheen MJC, Fuhler N, van Het Westeinde T, van der Pol CC, Young-Afat DA, Verkooijen HM. Compression Vest Treatment for Symptomatic Breast Edema in Women Treated for Breast Cancer: A Pilot Study. Lymphat Res Biol. 2020 Feb;18(1):56-63. doi: 10.1089/lrb.2018.0067. Epub 2019 Jun 18. PMID 31211631
- [Background] Verbelen H, De Vrieze T, Van Soom T, Meirte J, Van Goethem M, Hufkens G, Tjalma W, Gebruers N. Development and clinimetric properties of the Dutch Breast Edema Questionnaire (BrEQ-Dutch version) to diagnose the presence of breast edema in breast cancer patients. Qual Life Res. 2020 Feb;29(2):569-578. doi: 10.1007/s11136-019-02337-z. Epub 2019 Oct 28. PMID 31659592
- [Background] Mayrovitz HN, Somarriba C, Weingrad DN. Breast Tissue Dielectric Constant as a Potential Breast Edema Assessment Parameter. Lymphat Res Biol. 2022 Feb;20(1):33-38. doi: 10.1089/lrb.2020.0137. Epub 2021 Mar 24. PMID 33761280
- [Background] Kilbreath SL, Fearn NR, Dylke ES. Ultrasound: Assessment of breast dermal thickness: Reliability, responsiveness to change, and relationship to patient-reported outcomes. Skin Res Technol. 2022 Jan;28(1):111-118. doi: 10.1111/srt.13100. Epub 2021 Aug 29. PMID 34455642
- [Background] Yu Z, Liu N, Wang L, Chen J, Han L, Sun D. Assessment of Skin Properties in Chronic Lymphedema: Measurement of Skin Stiffness, Percentage Water Content, and Transepidermal Water Loss. Lymphat Res Biol. 2020 Jun;18(3):212-218. doi: 10.1089/lrb.2018.0066. Epub 2019 Oct 9. PMID 31596657
- [Background] Delay E, Gosset J, Toussoun G, Delaporte T, Delbaere M. [Post-treatment sequelae after breast cancer conservative surgery]. Ann Chir Plast Esthet. 2008 Apr;53(2):135-52. doi: 10.1016/j.anplas.2007.10.004. Epub 2008 Feb 20. French. PMID 18077074